CLINICAL TRIAL: NCT00510796
Title: A Pilot Study for Combined Colon and Endometrial Cancer Screening in Women at High-Risk for Colon and Endometrial Cancer
Brief Title: Combined Colon and Endometrial Cancer Screening in Women With HNPCC
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: ID01-694
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Colon Cancer
Keywords: Hereditary Non-Polyposis Colon Cancer; Colon Cancer; Endometrial Cancer; Cancer Screening; Interview; HNPCC
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis; Endometrial Neoplasms | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High Risk Group: Colon and/or Endometrial Cancer
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Interview regarding perception of pain and the benefits and barriers to the combined screening.
  Other Names: Survey

SUMMARY:
Primary Objectives:

To test the feasibility of combined colon and endometrial cancer screening in women with increased risk for colon and endometrial cancer.

To measure patient satisfaction for the combined procedure.

DETAILED DESCRIPTION:
Women with certain medical conditions have an increased risk for colon and endometrial cancer. Currently, women go through separate screening procedures. Endometrial biopsies are performed at a separate visit to the gynecologist, and patients are not sedated for the procedure. This study will involve performing an endometrial biopsy while you are sedated for your colonoscopy.

Women who are able to have children must have a negative blood or urine pregnancy test before they can take part in this study.

As part of the study, you will be asked about your past experience with endometrial biopsy and colonoscopy. You will be asked about your perception of pain, your expectations, and the benefits and barriers to the combined screening.

You will then be sedated. The colonoscopy will be performed first by a gastroenterologist. This will be followed by the endometrial biopsy, which will be performed by a gynecologic oncologist.

A telephone interview will be performed two weeks after this procedure. The interview will last about 15 minutes. You will be asked about your perception of pain and the benefits and barriers to the combined screening.

This is an investigational study. A total of 50 women will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1) Women with medical indications for colonoscopy and endometrial biopsy.

Exclusion Criteria:

1) Must be 18 years of age and older.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UT MDACC Female patients determined to be in a high risk group for either colon and/or endometrial cancer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2002-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Feasibility to perform both colon and endometrial cancer screening at the time of colonoscopy in women at high risk for colon and endometrial cancer. | 8 Years

CONTACTS AND LOCATIONS:
Overall Officials: Karen H. Lu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org